CLINICAL TRIAL: NCT04980560
Title: Longitudinal Assessment of Gut Microbiota Profile and Its Impact on Immunity Status in COVID-19 Vaccinated Cohorts in Hong Kong
Brief Title: Gut Microbiota Profile and Its Impact on Immunity Status in COVID-19 Vaccinated Cohorts
Status: Active, not recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Siew Chien NG, Professor, Chinese University of Hong Kong
Other Study IDs: MicVAC
Record Dates: First submitted 2021-07-26; First posted 2021-07-28 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: COVID-19 Vaccination; Gut Microbiota

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and stool samples will be collected
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- VAC cohort: Subjects who will take COVID-19 vaccines
- CON cohort: Subjects who are COVID-19 survivors

SUMMARY:
This study aims to examine the association between gut microbiota composition and the magnitude and duration of immune response in subjects who have received different COVID-19 vaccines in Hong Kong and to identify the differences compared to those COVID-19 recovered subjects.

DETAILED DESCRIPTION:
SARS-CoV-2, the cause of COVID-19, emerged as a new zoonotic pathogen of humans at the end of 2019 and rapidly developed into a global pandemic in March 2020. Over 106 million COVID-19 cases including 2.3 million deaths have been reported to the WHO as of February 9th 2021. Overall 80% of cases are mild/moderate or asymptomatic while 20% may develop severe or critical disease with respiratory failure requiring oxygen support and intensive care. As of 16 February 2021, 10789 cases have been confirmed in HK with 193 deaths while 10231 patients have been discharged from acute public hospitals with a mean length of stay of 15 days. Up to 16 Feb., 2021, there were 568 patients with COVID-19 have been managed at the Prince of Wales Hospital (PWH) with 12 deaths.

Studies showed that the quality of life of the patients who have recovered from COVID-19 was impaired. This situation is similar to some patients who suffered from SARS-CoV1 infection in 2003.

Natural infection by virus triggers an effective system immunity so that the host can resist or highly reduce the chance of re-infection.

In many cases, this protection can maintain a long period of time. On the other hand, vaccination, which aims to induce the similar immunity but in a controlled manner, presents only selected antigen(s) to the host through different delivery strategies. Lacking a normal virus replication cycle, vaccination can only partially mimic the infection process that makes the immunogenicity or durability of the vaccines sometimes not as effective as natural infection. This situation was also observed during the development of SARS and MERS vaccines. A number of studies focused on examining the humoral and cellular immunities from the COVID-19 patients during their acute stage or only few months after recovery. However, the long-term immunities (over a year) from the patients are not yet very clear.

The HKSAR government has procured 2 different types of COVID-19 vaccines for all the HK citizens that is one of the few regions/countries adopt this strategy. BioNTech mRNA vaccination programme will commence in early March 2021 and Sinovac inactivated whole virus vaccine will also be available soon for vaccination after formal approval recently. All these vaccines are so far only evaluated at their own designated population and countries and there is still lack of prospective study to "side-by-side" comparing the microbial biomarkers in the stool of different vaccines. Having different vaccines which will soon be available in Hong Kong, it would be of great interest to investigate and compare the microbial biomarkers in the stool of recovered COVID-19 patients versus those who have received different COVID-19 vaccines by setting up a 2-year longitudinal study.

ELIGIBILITY:
Inclusion Criteria for Vaccination (VAC) cohort:

1. aged ≥ 18 years old; and
2. have documented to have no previous COVID-19 infection; and
3. will receive any type of COVID-19 vaccines; and
4. agree to hand in study samples (stool and blood); and
5. agree to sign the informed consent

Inclusion Criteria for COVID-19 convalescent (CON) cohort:

1. aged ≥ 18 years old; and
2. recovered from varying severity of COVID-19; and
3. agree to hand in study samples (stool and blood); and
4. agree to sign the informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from different clinics in Prince of Wales Hospital, the CUHK Medical Centre, CUHK staff clinics, and community sources. Some subjects will be referred from other observational studies and some will be from any community source.
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To identify and compare the microbiome profile and immune response | 3 months
  To identify and compare the microbiome profile and immune response in subjects who have received different COVID-19 vaccines and in subjects who recovered from COVID-19 in Hong Kong

SECONDARY OUTCOMES:
SARS-CoV-2 IgG antibody level | across 24 months
  SARS-CoV-2 IgG antibody level in VAC cohort
Compare the serum neutralization assay against pseudovirus and live virus, as well as the detection of IgM and IgG against receptor-binding domain [RBD] and S1 | across 24 months
  Compare the serum neutralization assay against pseudovirus and live virus, as well as the detection of IgM and IgG against receptor-binding domain [RBD] and S1
SARS-CoV-2 specific antibody | across 24 months
  Compare the levels of SARS-CoV-2 specific antibody

CONTACTS AND LOCATIONS:
Overall Officials: Siew Ng, Principal Investigator — CUHK-M&T
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong